CLINICAL TRIAL: NCT06537934
Title: Advanced Mutidimensional and Ultra High Resolution Computed Tomography to Inspect Cardiopulmonary Involvement in Progressive Fibrosing Interstitial Lung Diseases
Acronym: AMICI-ILD
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Anna Palmisano, Professor, IRCCS San Raffaele
Other Study IDs: PNRR-MCNT2- 2023-12377844
Record Dates: First submitted 2024-06-10; First posted 2024-08-05 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Diseases
Keywords: Cardiac fibrosis; Lung interstitial fibrosis
MeSH Terms: conditions — Lung Diseases, Interstitial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Interstitial lung diseases (ILDs) are common chronic disease characterized by high mortality and morbidity, also linked to cardiovascular implication. Cardiovascular complications, occur early in idiopathic pulmonary fibrosis (IPF) and other ILDs without anysymptoms. Symptoms are often misinterpreted and diagnosis delayed to irreversible stages of cardiac dysfunction. Mechanism of cardiac damage, the main cause of mortality, are heterogeneous raging from ischemic heart disease, acceleration of atherosclerosis, to right ventricle dysfunction secondary, to pulmonary hypertension. So an early recognition and accurate staging are fundamental to avoid disease progression and improve outcomes. The identification of a single non-invasive imaging modality able to simultaneously characterize in an accurate and quantitative way the entity of lung and cardiac damage in patients affected by ILD would be useful to improve risk stratification and to guide treatment.

ELIGIBILITY:
Inclusion Criteria:

• Adult subjects (>18 y.o.) with previously known ILD or high likelihood for having ILD including CTD diagnosis since at least 5 years before the project starts in order to increase the prevalence of ILD [2] who signed an Informed Consent authorizing data collection.

Exclusion Criteria:

* Subjects with active infectious disease;
* known CAD;
* history of previous percutaneous or surgical revascularization;
* known cardiomyopathy;
* previous heart failure;
* presence of cardiac devices (prosthetic valve, ICD, PM, ICD-CRT, LVAD)
* previous or active neoplasia;
* pregnancy and breastfeeding;
* allergy to iodine contrast agent;
* claustrophobia;
* glomerular filtration rate < 30mL/min
* impossibility to lay down or breath old
* absence of informed consent signed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 123 patients will be submitted to standard of care imaging and the informed consent is required for the authorization to use the imaging data for scientific purpose and to collected clinical and laboratory data using electronic medical records, and clinical interview.
  All patients will undergo echocardiography, as clinically indicated, that will be performed in accordance with the most recent guidelines for a comprehensive morphofuctional assessment of cardiac chambers, valves, evaluation of pulmonary hypertension and associated remodeling, including the identification of subtle myocardial deformation alteration using strain analysis. Hence, CT will be compared to echocardiography, currently indicated for the monitoring of CTD, in order to establish agreement and potential additional information. Hence, only a subgroup of 74 patients who have an altered troponin T value (> 14 ng/L) will undergo cardiac magnetic resonance imaging (CMR) according to clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 123 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-09-01 (Actual); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
a low dose image protocol able to characterize ILD related lung parenchyma alteration and new quantitative imaging biomarkers of lung disease severity | months 2-12

SECONDARY OUTCOMES:
the prevalence and the spectrum of cardiac disease (ischemic heart disease, cardiac remodelling and dysfunction in patients with ILD) and the relationship between severity of lung involvement and cardiac injury | months 3-16
a CT based multiparametric algorithm for risk stratification of patients with ILD | months 19-24

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS San Raffaele, Milan, Italy

REFERENCES:
- [Background] Wells AU, Brown KK, Flaherty KR, Kolb M, Thannickal VJ; IPF Consensus Working Group. What's in a name? That which we call IPF, by any other name would act the same. Eur Respir J. 2018 May 17;51(5):1800692. doi: 10.1183/13993003.00692-2018. Print 2018 May. PMID 29773608
- [Background] Sauleda J, Nunez B, Sala E, Soriano JB. Idiopathic Pulmonary Fibrosis: Epidemiology, Natural History, Phenotypes. Med Sci (Basel). 2018 Nov 29;6(4):110. doi: 10.3390/medsci6040110. PMID 30501130
- [Background] Gupta S, Padhan P, Subhankar S, Singh P. Cardiovascular complications in patients with interstitial lung disease and their correlation with 6-minute walk test and spirometry: A single-center study. J Family Med Prim Care. 2021 Sep;10(9):3330-3335. doi: 10.4103/jfmpc.jfmpc_350_21. Epub 2021 Sep 30. PMID 34760753
- [Background] Raghu G, Amatto VC, Behr J, Stowasser S. Comorbidities in idiopathic pulmonary fibrosis patients: a systematic literature review. Eur Respir J. 2015 Oct;46(4):1113-30. doi: 10.1183/13993003.02316-2014. PMID 26424523
- [Background] Raghu G, Remy-Jardin M, Myers JL, Richeldi L, Ryerson CJ, Lederer DJ, Behr J, Cottin V, Danoff SK, Morell F, Flaherty KR, Wells A, Martinez FJ, Azuma A, Bice TJ, Bouros D, Brown KK, Collard HR, Duggal A, Galvin L, Inoue Y, Jenkins RG, Johkoh T, Kazerooni EA, Kitaichi M, Knight SL, Mansour G, Nicholson AG, Pipavath SNJ, Buendia-Roldan I, Selman M, Travis WD, Walsh S, Wilson KC; American Thoracic Society, European Respiratory Society, Japanese Respiratory Society, and Latin American Thoracic Society. Diagnosis of Idiopathic Pulmonary Fibrosis. An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline. Am J Respir Crit Care Med. 2018 Sep 1;198(5):e44-e68. doi: 10.1164/rccm.201807-1255ST. PMID 30168753
- [Background] Gaillandre Y, Duhamel A, Flohr T, Faivre JB, Khung S, Hutt A, Felloni P, Remy J, Remy-Jardin M. Ultra-high resolution CT imaging of interstitial lung disease: impact of photon-counting CT in 112 patients. Eur Radiol. 2023 Aug;33(8):5528-5539. doi: 10.1007/s00330-023-09616-x. Epub 2023 Apr 18. PMID 37071165
- [Background] Palmisano A, Vignale D, Tadic M, Moroni F, De Stefano D, Gatti M, Boccia E, Faletti R, Oppizzi M, Peretto G, Slavich M, Sala S, Montorfano M, Agricola E, Margonato A, De Cobelli F, Gentile F, Robella M, Cortese G, Esposito A. Myocardial Late Contrast Enhancement CT in Troponin-Positive Acute Chest Pain Syndrome. Radiology. 2022 Mar;302(3):545-553. doi: 10.1148/radiol.211288. Epub 2021 Dec 7. PMID 34874200
- [Background] Vignale D, Palmisano A, Colantoni C, Brunetti L, Nicoletti V, Gnasso C, Esposito A. Toward a One-Stop Shop CT Protocol in Acute Chest Pain Syndrome. Radiology. 2023 Jan;306(1):E3-E4. doi: 10.1148/radiol.220844. Epub 2022 Sep 27. No abstract available. PMID 36165795
- [Background] Palmisano A, Gnasso C, Cereda A, Vignale D, Leone R, Nicoletti V, Barbieri S, Toselli M, Giannini F, Loffi M, Patelli G, Monello A, Iannopollo G, Ippolito D, Mancini EM, Pontone G, Vignali L, Scarnecchia E, Iannaccone M, Baffoni L, Spernadio M, de Carlini CC, Sironi S, Rapezzi C, Esposito A. Chest CT opportunistic biomarkers for phenotyping high-risk COVID-19 patients: a retrospective multicentre study. Eur Radiol. 2023 Nov;33(11):7756-7768. doi: 10.1007/s00330-023-09702-0. Epub 2023 May 11. PMID 37166497
- [Background] Pontone G, Baggiano A, Conte E, Teruzzi G, Cosentino N, Campodonico J, Rabbat MG, Assanelli E, Palmisano A, Esposito A, Trabattoni D. "Quadruple Rule-Out" With Computed Tomography in a COVID-19 Patient With Equivocal Acute Coronary Syndrome Presentation. JACC Cardiovasc Imaging. 2020 Aug;13(8):1854-1856. doi: 10.1016/j.jcmg.2020.04.012. Epub 2020 Apr 21. No abstract available. PMID 32762888